CLINICAL TRIAL: NCT00112697
Title: Randomized Phase II Trial Evaluating [Radiotherapy-Docetaxel-5 Fluorouracil] Association Versus [Radiotherapy-Docetaxel-Cisplatin] Association in Non Resecables First Line of Chemotherapy in Metastatics Pancreas Cancers Patients
Brief Title: Radiation Therapy and Docetaxel With Either Fluorouracil or Cisplatin as First-Line Therapy in Treating Patients With Metastatic Pancreatic Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000430095; FRE-FNCLCC-ACCORD-09/0201; EU-20511
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cisplatin; Docetaxel; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: docetaxel; Drug: fluorouracil; Radiation: radiation therapy
- Arm 2 (Experimental)
  Interventions: Drug: cisplatin; Drug: docetaxel; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
  Arms: Arm 2
Drug: docetaxel
Drug: fluorouracil
  Arms: Arm 1
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as docetaxel, fluorouracil, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with chemotherapy may kill more tumor cells. It is not yet known whether radiation therapy, docetaxel, and fluorouracil are more effective than radiation therapy, docetaxel, and cisplatin as first-line therapy in treating pancreatic cancer.

PURPOSE: This randomized phase II trial is studying radiation therapy, docetaxel, and fluorouracil to see how well they work as first-line therapy compared to radiation therapy, docetaxel, and cisplatin in treating patients with metastatic pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the 6-month progression-free survival rate in patients with unresectable metastatic adenocarcinoma of the pancreas treated with radiotherapy and docetaxel in combination with either fluorouracil or cisplatin as first-line therapy.

Secondary

* Compare the toxicity of these regimens in these patients.
* Compare the objective response rate in patients treated with these regimens.
* Compare overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radiotherapy to the celiac area once daily 5 days a week for 6 weeks. Patients also receive docetaxel IV weekly and fluorouracil IV daily for 6 weeks.
* Arm II: Patients undergo radiotherapy and receive docetaxel as in arm I. Patients also receive cisplatin IV weekly for 6 weeks.

In both arms, patients experiencing disease progression after completion of chemoradiotherapy may receive additional courses of chemotherapy.

PROJECTED ACCRUAL: A total of 80 patients (40 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * No other pancreatic tumor type, including either of the following:

    * Neuroendocrine tumor
    * Ampulla of Vater carcinoma
  * Metastatic disease
* Measurable or evaluable disease
* Unresectable disease, defined as either of the following:

  * Failed prior attempt of surgical resection by laparotomy
  * Surgical resection contraindicated by radiographic criteria (e.g., arterial vascular invasion)
* No cerebral metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin < 1.5 times upper limit of normal
* No hepatic disturbance

Renal

* Creatinine < 120 mmol/L

Cardiovascular

* No untreated cardiac or coronary insufficiency
* No uncontrolled symptomatic arrhythmia
* No uncontrolled angina

Pulmonary

* No uncontrolled respiratory insufficiency

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* No peripheral neuropathy ≥ grade 2
* No ongoing active infection
* No other serious uncontrolled medical disorder that would preclude study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the celiac or pancreatic area

Surgery

* See Disease Characteristics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2003-10-06 (Actual); Primary Completion 2008-08-01 (Actual); Study Completion 2012-03-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate at 6 months

SECONDARY OUTCOMES:
Toxicity
Objective response rate
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Michel Ducreux, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (10):
- France (10):
  - Centre Paul Papin, Angers
  - Centre Oscar Lambret, Lille
  - Polyclinique des Quatre Pavillons, Lormont
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Oberic L, Viret F, Baey C, Ychou M, Bennouna J, Adenis A, Peiffert D, Mornex F, Pignon JP, Celier P, Berille J, Ducreux M. Docetaxel- and 5-FU-concurrent radiotherapy in patients presenting unresectable locally advanced pancreatic cancer: a FNCLCC-ACCORD/0201 randomized phase II trial's pre-planned analysis and case report of a 5.5-year disease-free survival. Radiat Oncol. 2011 Sep 26;6:124. doi: 10.1186/1748-717X-6-124. PMID 21943032